CLINICAL TRIAL: NCT00012155
Title: A Phase I, Open-Label, Dose-Escalating Study Of The Safety, Tolerability, And Anti-Tumor Activity Of A Single Intrahepatic Arterial Injection Of Genetically Engineered Herpes Simplex Virus, NV1020, In Subjects With Adenocarcinoma Of The Colon With Metastasis To The Liver
Brief Title: Gene Therapy in Treating Patients With Colon Cancer That Has Spread to the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-00022; CDR0000068488 (Registry Identifier: PDQ (Physician Data Query)); MGENE-NR1-001; NCI-G01-1920
Record Dates: First submitted 2001-03-03; First posted 2003-06-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2002-11

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; recurrent colon cancer; adenocarcinoma of the colon; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms

INTERVENTIONS:
Biological: NV1020

SUMMARY:
RATIONALE: Gene therapy may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the safety of NV1020 in patients who have colon cancer that has spread to the liver and has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and maximum tolerated dose of a single intrahepatic NV1020 injection in patients with hepatic metastases from colon cancer that has failed first-line chemotherapy.
* Determine the tolerability of this drug in these patients.
* Determine preliminarily the anti-tumor activity of this drug in these patients.
* Assess the immunogenicity of NV1020 in these patients.

OUTLINE: This is a dose escalation study.

Patients receive a single intrahepatic arterial injection of NV1020 over 10 minutes with the aid of hepatic arteriography.

Cohorts of 3 patients receive escalating doses of NV1020 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity.

Patients are followed at 1, 2, and 3 months post injection. Patients may participate in a separate long term (up to 1 year) follow-up study for continued assessment and monitoring.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon

  * At least 3 metastatic hepatic lesions involving both lobes
  * No extrahepatic disease
* Failed first-line combination chemotherapy of fluorouracil plus either leucovorin calcium or irinotecan
* Herpes simplex virus type-1 seropositive
* Candidate for intrahepatic arterial infusion pump placement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9.0 g/dL
* No history of any blood clotting disorder (e.g., hemophilia)

Hepatic:

* Transaminases no greater than 3 times upper limit of normal
* Bilirubin no greater than 2.0 mg/dL
* No active hepatitis
* No history of hepatic fibrosis, cirrhosis, or hemochromatosis

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* All patients must use effective barrier contraception during and for at least 6 months after study
* HIV negative
* No active herpes infection
* No other active uncontrolled infection
* No prior weight loss of more than 10 lbs within the past month
* No history of alcohol or other substance abuse
* No concurrent unstable and/or severe medical or psychological condition
* No history of any other medical or psychological condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy (e.g., interleukin-2, interleukin -12, or interferon)
* No prior gene transfer therapy
* No prior therapy with cytolytic virus of any type
* No concurrent immunotherapy during and for 28 days after study therapy
* No concurrent vaccines during and for 28 days after study therapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy during and for 28 days after study therapy

Endocrine therapy:

* No concurrent systemic steroids during and for 28 days after study therapy

Radiotherapy:

* No prior radiotherapy to the liver
* No concurrent radiotherapy during and for 28 days after study therapy

Surgery:

* At least 2 weeks since prior surgery

Other:

* At least 30 days since prior participation in investigational study
* No concurrent antiviral agent active against herpes simplex virus (e.g., acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, or cidofovir) during and for 28 days after study therapy
* No concurrent immunosuppressive agents (e.g., cyclosporine) during and for 28 days after study therapy
* No other concurrent investigational or anti-cancer agents during and for 28 days after study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2002-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuman Fong, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kemeny N, Jarnagin W, Guilfoyle B, et al.: Results of a phase I, dose-escalating study of the safety, tolerability and anti-tumor activity of a single injection of a genetically engineered herpes simplex virus, nv1020, in subjects with hepatic colorectal metastases. [Abstract] Ann Oncol 16 (Suppl 2): A-480, ii283, 2005.